CLINICAL TRIAL: NCT02756507
Title: The Efficacy of a Video-based Transdiagnostic REBT Universal Prevention Program Delivered in a School Context for Internalizing Problems in Adolescents
Brief Title: Transdiagnostic REBT Prevention Program for Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Anca Dobrean, Ph.D., Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PN-II-PT-PCCA-2011-3.1-1500
Record Dates: First submitted 2016-04-25; First posted 2016-04-29 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Social Anxiety; Major Depression Mild; Panic Disorder; Specific Phobia; Generalized Anxiety Disorder
Keywords: anxiety symptoms; depression symptoms; internalizing symptoms
MeSH Terms: conditions — Panic Disorder; Phobia, Specific; Generalized Anxiety Disorder; Anxiety Disorders; Depression | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- video-based transdiagnostic REBT (Experimental): Children and adolescents in the experimental group attend 6 modules of video-based transdiagnostic rational emotive behavioral therapy (REBT). Each of the six modules aimes a different component: Psychoeducation, Relaxation, Relationship between cognitive distortions/irrational beliefs and emotions, Cognitive restructuring, Exposure/ behavior activation and problem solving, Maintenance of gaining.
  Interventions: Behavioral: video-based transdiagnostic REBT
- wait list (Sham Comparator): The wait-list is a delayed treatment condition.
  Interventions: Behavioral: Wait list

INTERVENTIONS:
Behavioral: video-based transdiagnostic REBT — The video-based transdiagnostic REBT consists of 6 sessions delivered in a group format.
  Arms: video-based transdiagnostic REBT
Behavioral: Wait list — Delayed intervention
  Arms: wait list

SUMMARY:
Anxiety and depressive disorders are common in adolescents, however they are often unrecognized. Rational emotive behavioral therapy (REBT), a form of cognitive behavioral therapy (CBT) is efficient for children and adolescents. School settings are appropriate environments to deliver such interventions for vulnerable youths. Given youth's access and predilection to use technology, a video-based prevention program was developed. The present study aims to investigate the efficacy of a transdiagnostic REBT prevention program for internalizing symptoms in adolescents, implemented in a school setting.

Classes from different Romanian public schools will be randomized in either intervention or wait list group.

DETAILED DESCRIPTION:
The prevention program will be group-based, delivered in 6 sessions, over 3 weeks.

Each of the six modules aimed a different component: Psychoeducation, Relaxation, Relationship between cognitive distortions/irrational beliefs and emotions, Cognitive restructuring, Exposure/ behavioral activation and problem solving, Maintenance of gainings. Despite specific activities, for each session a video cartoon on that subject will be viewed and discussed. Homework would be given at every session.

REBT prevention programs delivered in school settings represent ecological modalities to target vulnerable groups. Technology components added to traditional programs may lead to greater motivation and satisfaction with treatment.

Adolescents will complete assessments at four time-points: T1 (baseline), T2 (post-intervention), T3 (3 months follow-up) and T4 (12 months follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Preadolescents and adolescents will have ages between 12 and 17 years old;
2. Are attending middle school or high-school;
3. Adolescents have sufficient understanding of the Romanian language in order to complete assessments at all time points and to participate in the prevention program;
4. Their parents have sufficient understanding of the Romanian language in order to sign the informed consent;
5. Parents will sign the informed consent and adolescents will provide informed assent.

Exclusion Criteria:

1. Age below 14 or above 17 years;
2. No signed informed consent from parents;
3. Adolescents will score high on suicidal ideation according to (1 item on the Depression subscale from Beck Youth Inventories);
4. Not Romanian-speaking in order to understand the content of the prevention program and to complete the assessments.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 381 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
The Multidimensional Anxiety Scale for Children (MASC; March, Parker, Sullivan, Stallings, & Conners, 1997) | Change from baseline anxiety symptoms at 3 weeks post-intervention, 3 months follow up, 12 months follow-up
  anxiety symptoms
Beck Depression Inventory for Youth subscale from the Beck Youth Inventories-Second edition for children and adolescents (Beck, 2005) | Change from baseline depressive symptoms at 3 weeks post-intervention, 3 months follow up, 12 months follow-up
  depressive symptoms

SECONDARY OUTCOMES:
The Children's Automatic Thoughts Scale - Negative/Positive (CATS-N/P) (Hogendoorn et al., 2010) | Change from baseline maladaptive cognitions at 3 weeks post-intervention, 3 month follow up, 12 months follow-up
  maladaptive cognitions
The Strengths and Difficulties Questionnaire (SDQ) (Goodman, 1997) | Change from baseline comorbid problems at 3 weeks post-intervention, 3 months follow up, 12 months follow-up
  comorbid problems
The Questionnaire for Measuring Health-Related Quality of Life in Children and Adolescents, The Revised Version - adolescent version (Kiddo-KINDL) (Ravens-Sieberer et al., 2001) | Change from baseline quality of life at 3 weeks post-intervention, 3 months follow up, 12 months follow-up
  quality of life
The Credibility/ Expectancy Questionnaire (Devilly & Borkovec, 2000) | pre-intervention
  Treatment expectancies
The Client Satisfaction Scale (Vigerland et al., 2016) | post-intervention
  Satisfaction with the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Anca Dobrean, Ph.D., Study Director — Babes-Bolyai University
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be shared upon reasonable request after the publication of the manuscripts resulting from this study.
Access Criteria: Data will be requested from the corresponding author of the resulting papers.

REFERENCES:
- [Derived] Pasarelu CR, Dobrean A. A video-based transdiagnostic REBT universal prevention program for internalizing problems in adolescents: study protocol of a cluster randomized controlled trial. BMC Psychiatry. 2018 Apr 13;18(1):101. doi: 10.1186/s12888-018-1684-0. PMID 29653523